CLINICAL TRIAL: NCT06124092
Title: After Pediatric Critical Illness (APCI)
Brief Title: Outcomes of Children After Hospitalization in Intensive Care Unit
Acronym: APCI
Status: Not yet recruiting | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Genevieve Du Pont-Thibodeau, MD, St. Justine's Hospital
Other Study IDs: CHUSJ MP-21-2023-5097
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Renal Disease; Liver Diseases; Heart Diseases; Trauma Injury; Sepsis; Septic Shock; Pneumonia; Bronchiolitis
Keywords: Pediatric Intensive Care Unit; PICU
MeSH Terms: conditions — Kidney Diseases; Liver Diseases; Heart Diseases; Accidental Injuries; Sepsis; Shock, Septic; Pneumonia; Bronchiolitis | interventions — Mental Status and Dementia Tests; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: neurocognitive tests — Cohort study: all parents and participants will have questionnaires to complete, based on participant's age.
  Other Names: Quality of life

SUMMARY:
More than 10,000 children are hospitalized in an PICU every year in Canada. While most of them will survive their PICU hospitalization and their critical illness, some children will not recover to their pre-illness level. Some may develop behavioral, physical, emotional or developmental problems and difficulties at school. All these problems are elements that are part of the Pediatric Post-Intensive Care Syndrome (PICS-p).

It is important to understand the elements (risk factors) that play a role in the development of PICS-p. In Canada, there is no systematic follow-up for children after they leave the PICU. Understanding what can cause PICS-p (risk factors) and how much PICS-p has an impact on children and their family is very important to the family well-being.

DETAILED DESCRIPTION:
The Pediatric Post-Intensive Care Syndrome (PICS-p) is a newly developed conceptual framework that incorporates the constellation of morbidities that are increasingly recognized to affect children and their families after a critical illness. Experts define PICS-p as a new or worsening impairment in any of the following 5 domains of child health: physical, cognitive, emotional, social, or family.

In contrast to well established follow-up programs in adults, there is currently a lack of systematic follow-up of PICU survivors which prevents both the recognition and management of PICS-p. The absence of granular, empirical data on the recovery of PICU children impedes both the identification and management of PICS-p.

This project is a prospective Canadian multicenter cohort study to identify risk factors of PICS-p, develop and validate a predictive model for PICS-p to detect at-risk children, characterize each domain of PICS-p over two years post critical illness and uncover additional morbidities that are not captured using the current PICS-p framework. This study will provide granular, empirical data on which to build developmentally appropriate and tailored screening, management, and intervention programs during and after PICU to improve the global recovery of critically ill children and their family.

ELIGIBILITY:
Inclusion Criteria:

* Children ≤18yo hospitalized in PICU for ≥96 hours

Exclusion Criteria:

1. gestational age <37 weeks or age >18 years at PICU entry;
2. admitted for congenital heart surgery (followed in neuro-cardiac clinics in most centers);
3. anticipated life expectancy <1year (e.g., active do not resuscitate status).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient admitted to Pediatric Intensive Care Unit for 96 hours or more will be included in the study unless they age a gestionnal age <37 weeks or are over 18 years-old or were admitted to PICu for congenital heart surgery (as they are followed in neuro-cardiac clinic) and for whom the life expectancy is less than 1 year.
Sampling Method: Probability Sample
Enrollment: 690 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Identify risk factors of PICS-p at 2 months post-PICU | 2 months after PICU discharge
  Identification of modifiable and non-modifiable risk factors
Develop and validate a model predictive of PICS-p 2 months post PICU | 2 months after PICU discharge
  The model will allow detection at PICU discharge of children in need of post-PICU follow-up

SECONDARY OUTCOMES:
Describe the incidence of each of the five domains of PICS-p across the first two years post-PICU | At 2 months, 12, 18 months and 36 months post PICU discharge
  Identify which domain gets impacted and when during the course of the follow-up
Uncover additional post-PICU morbidities not detected within the framework of PICS-p. | Until 36 months post PICU discharge
  Detection of morbidities through the medical provider interview that are not included in the current framework.

OTHER OUTCOMES:
Describe families' healthcare requirements throughout their recovery process after PICU. | Until 36 months post PICU discharge
  Descrie the variety of healthcare professional and medical required post PICU hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève Du Pont-Thibodeau, MD, Principal Investigator — St. Justine's Hospital; Laurence Cucharme-Crevier, MD, Principal Investigator — St. Justine's Hospital
Locations (8):
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children Hospital, Vancouver, British Colombia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Childrens Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - Montreal Children Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided